CLINICAL TRIAL: NCT05748067
Title: Outcome of Minimally Invasive Treatment for Permanent Molars Affected With Molar-incisor Hypomineralization Defects: a Randomized Clinical Trial
Brief Title: Minimally Invasive Treatment for Permanent Molars Affected With Molar-incisor Hypomineralization Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 623-2021
Record Dates: First submitted 2023-02-05; First posted 2023-02-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: SDF, HVGIC & SSC (Active Comparator): Silver diamine fluoride (SDF) will be clinically applied in the first visit. After 1 week of caries arrest, the tooth will be restored with a high viscosity glass ionomer (HVGIC) and stainless steel crown (SSC).
  Interventions: Procedure: SDF; Procedure: HVGIC restoration; Procedure: SSC
- Group 2: SDF & SSC (Active Comparator): Silver diamine fluoride (SDF) will be clinically applied in the first visit. After 1 week of caries arrest, the tooth will be restored with a SSC only.
  Interventions: Procedure: SDF; Procedure: SSC
- Group 3: HVGIC & SSC (Active Comparator): The tooth will be restored in a similar fashion to atraumatic restorative treatment (ART technique) and restored with a high viscosity glass ionomer (HVGIC) and stainless steel crown (SSC).
  Interventions: Procedure: HVGIC restoration; Procedure: SSC

INTERVENTIONS:
Procedure: SDF — Silver diamine fluoride
  Arms: Group 1: SDF, HVGIC & SSC; Group 2: SDF & SSC
Procedure: HVGIC restoration — High viscosity glass ionomer restoration
  Arms: Group 1: SDF, HVGIC & SSC; Group 3: HVGIC & SSC
Procedure: SSC — Stainless steel crown

SUMMARY:
In this prospective randomized clinical trial, the is aim to compare the clinical and radiographic success of 3 minimally invasive treatment protocols on permanent first molars affected with MIH over 24 months. A total of 73children/120molar teeth (N=40 molars per group) between the ages of 6-16 years with MIH will be recruited at the post-graduate clinics at Jordan University of Science and Technology (JUST).

DETAILED DESCRIPTION:
Background: The term molar-incisor hypomineralization (MIH) is defined as 'hypomineralization of systemic origin, presenting as demarcated, qualitative defects of enamel of one to four first permanent molars (FPMs) frequently associated with affected incisors. There are no clinical studies on use of minimally invasive techniques as restorative treatments for molars affected by MIH.

Aim: The aim of this clinical trial is to compare the clinical and radiographic success of 3 minimally invasive treatment protocols on permanent first molars affected with MIH over 24 months.

Methods: A total of 73 children/120 molar teeth (N=40 molars per group) between the ages of 6-16 years with MIH will be recruited for this prospective randomized clinical trial in the post-graduate clinics at JUST. Clinical and radiographic examination will be done. Participants will be randomly allocated to one of the three treatment modalities: For groups 1 and 2, silver diamine fluoride (SDF) will be clinically applied using cotton roll isolation on the first visit for three minutes after cleaning the tooth with gauze. After 1 week, the carious lesion will be examined for signs of caries arrest using two criteria: the color turning darker black and increased hardness of the lesion rather than soft texture (assessed using an excavator), if the criteria are met, the tooth will be restored with high viscosity glass ionomer (HVGIC) and stainless steel crown (SSC) for group 1, or only with a SCC for group 2. If not met, the carious lesion will be assumed to be still active, and a reapplication of SDF will be done before restoring the tooth with HVGIC and SCC. In group 3, the tooth will be restored in a similar fashion to atraumatic restorative treatment (ART technique) and restored with HVGIC and a SCC. Follow up will be done for all groups at 3 months, 6 months, 12 months, and 24 months to record specified clinical and radiographic criteria as outcome measures of success.

ELIGIBILITY:
Inclusion Criteria:

* Permanent molars with MIH with the following MIH indices (2a, 2b, 3, 4a, 4b) affected by caries (ICDAS 3 or 4) or post eruptive breakdown.
* Restorable teeth
* Permanent molars with MIH with NO clinical/radiographic signs and symptoms of irreversible pulpitis or pulpal necrosis.
* Clear band of dentine radiographically between the carious lesion and the pulp.

Exclusion Criteria:

* Medically compromised patients.
* Permanent molars with MIH with the following indices (1, 2c, 4c, 0, 1).
* Permanent molars with MIH with severe post eruptive breakdown therefore, unrestorable.
* Permanent molars with MIH with clinical/radiographic signs and symptoms of irreversible pulpitis or pulpal necrosis.
* No clear band of dentine radiographically between the carious lesion and the pulp.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Successful restoration | After 1 year
  SSC is clinically intact (not perforated), retentive (not lost), in proper occlusion, with no gingival inflammation
Functional tooth clinically | After 1 year
  Tooth should have no symptoms of pain, mobility or tenderness to percussion
Healthy periapical region radiographically | After 1 year
  No signs of periapical pathology on radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Ola B. Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghanim A, Silva MJ, Elfrink MEC, Lygidakis NA, Marino RJ, Weerheijm KL, Manton DJ. Molar incisor hypomineralisation (MIH) training manual for clinical field surveys and practice. Eur Arch Paediatr Dent. 2017 Aug;18(4):225-242. doi: 10.1007/s40368-017-0293-9. Epub 2017 Jul 18. PMID 28721667
- [Background] Ozgul BM, Saat S, Sonmez H, Oz FT. Clinical evaluation of desensitizing treatment for incisor teeth affected by molar-incisor hypomineralization. J Clin Pediatr Dent. 2013 Winter;38(2):101-5. PMID 24683770
- [Background] Steffen R, Kramer N, Bekes K. The Wurzburg MIH concept: the MIH treatment need index (MIH TNI) : A new index to assess and plan treatment in patients with molar incisior hypomineralisation (MIH). Eur Arch Paediatr Dent. 2017 Oct;18(5):355-361. doi: 10.1007/s40368-017-0301-0. Epub 2017 Sep 14. PMID 28913739
- [Background] Jalevik B, Klingberg GA. Dental treatment, dental fear and behaviour management problems in children with severe enamel hypomineralization of their permanent first molars. Int J Paediatr Dent. 2002 Jan;12(1):24-32. PMID 11853245
- [Background] Zhao IS, Gao SS, Hiraishi N, Burrow MF, Duangthip D, Mei ML, Lo EC, Chu CH. Mechanisms of silver diamine fluoride on arresting caries: a literature review. Int Dent J. 2018 Apr;68(2):67-76. doi: 10.1111/idj.12320. Epub 2017 May 21. PMID 28542863
- [Background] Grossi JA, Cabral RN, Ribeiro APD, Leal SC. Glass hybrid restorations as an alternative for restoring hypomineralized molars in the ART model. BMC Oral Health. 2018 Apr 18;18(1):65. doi: 10.1186/s12903-018-0528-0. PMID 29669561
- [Background] Horst JA, Ellenikiotis H, Milgrom PL. UCSF Protocol for Caries Arrest Using Silver Diamine Fluoride: Rationale, Indications and Consent. J Calif Dent Assoc. 2016 Jan;44(1):16-28. PMID 26897901
- [Background] Crystal YO, Marghalani AA, Ureles SD, Wright JT, Sulyanto R, Divaris K, Fontana M, Graham L. Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. Pediatr Dent. 2017 Sep 15;39(5):135-145. PMID 29070149